CLINICAL TRIAL: NCT00573365
Title: LED Photomodulation for Prevention of Post-Radiation Treatment Dermatitis: A Prospective, Randomized, Controlled Study
Brief Title: LED Photomodulation for Prevention of Post-Radiation Treatment Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: UCI 06-46; 2006-5251 (Other: University of California, Irvine)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Radiation Dermatitis
Keywords: dermatitis; skin; radiation; light; LED photomodulation; Gentlewaves
MeSH Terms: conditions — Radiodermatitis; Dermatitis | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: The enrollment goal of 40 includes 20 for each arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): LED treatment with Gentlewaves Select™ handheld high energy LED array 5 to 10 minutes before each radiation treatment and again 5-10 minutes after each radiation treatment
  Interventions: Device: Gentlewaves Select™ handheld high energy LED array; Radiation: Radiation
- Control (Other): Radiation only
  Interventions: Radiation: Radiation

INTERVENTIONS:
Device: Gentlewaves Select™ handheld high energy LED array — LED photomodulation within 5-10 minutes before and within 5-10 minutes after each radiation treatment
  Arms: Treatment
Radiation: Radiation — Weekly radiation treatment
  Arms: Control
Radiation: Radiation — Weekly radiation treatment
  Arms: Treatment

SUMMARY:
Radiation dermatitis is a common side-effect of radiation therapy in cancer patients who frequently can experience redness, pain, crusting, and even ulceration of the skin causing suffering and treatment interruption. A recent retrospective study by DeLand demonstrated that administering light emitting diode (LED) photomodulation after each radiation treatment for breast cancer decreased radiation dermatitis in a majority of patients. LED photomodulation is a process by which specific sequences of light are used to regulate or manipulate cell activity without causing heat or damage to the skin. Each LED treatment is painless and is completed in usually less than one minute. LED photomodulation may reduce the suffering associated with radiation treatments, improve cosmetic outcome in radiation fields, and eliminate breaks in radiation treatments which may be required because of severe ulcerating reactions.

This study will attempt to replicate the findings of Dr. DeLand's study by randomly assigning at least 40 breast cancer patients to either a treatment group or to a control group. The treatment group will receive LED photomodulation treatments before and after each radiation treatment with the Gentlewaves Select™ handheld high energy 590nm LED array using specific sequences of pulses used in other studies; the treatment group will also receive 7 additional treatments over 2 weeks after their radiation treatment course is completed. The control group will receive no LED treatment but will use the exact same skin care regimen as the treatment group. In addition to weekly evaluation and grading of skin reactions, subjects will be photographed under standardized conditions weekly and then photographs will be evaluated and graded by blinded dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clinically diagnosed breast or head and neck cancer that will be treated with radiation therapy.
* Subjects must be at least 18 years of age

Exclusion Criteria:

* Subjects will not be eligible to participate if they are pregnant or lactating.
* Patients treated with partial breast irradiation techniques, brachytherapy, or other non-standard techniques will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Determine efficacy | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Fife, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States